CLINICAL TRIAL: NCT00294788
Title: Phase I/II Placebo-Controlled Study of Consumption of a Probiotic on HAI Titre Following Influenza Vaccination of Healthy Adult Subjects
Brief Title: Evaluation of the Safety and Effectiveness of a Probiotic Bacterium to Boost the Immune Response to Influenza Vaccines
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Probiomics Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ProFlu2006; H05/123
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Influenza
Keywords: Influenza; bioadjuvant; probiotic; HAI; immunity; vaccine; Immune response to influenza vaccine
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: Fluvax
Drug: PCC® (Lactobacillus fermentum VRI 003)

SUMMARY:
This project aims to test the hypothesis that oral consumption of a specific strain of the probiotic bacterium Lactobacillus fermentum (trademarked PCC®) is able to significantly enhance the immune response to a vaccine for influenza.

ELIGIBILITY:
Inclusion Criteria:

* Persons must be adult men and women aged 18-49 years (have not reached 50th birthday).
* Persons must be able and willing to provide informed consent.
* Persons must be willing to receive the influenza vaccine (Fluvax®) given as an intramuscular injection.
* Persons must be willing to consume one gelatin capsule per day containing either probiotic bacteria or placebo (inactive substance) for the duration (42 days) of the study.
* Persons must be willing to provide blood specimens, each of 10 ml, collected by venepuncture.
* Persons must be willing to notify study personnel of a range of health effects by questionnaire.

Exclusion Criteria:

* Any health condition for which the influenza vaccine is not recommended including: chronic diseases of the pulmonary or cardiovascular systems (including asthma); chronic metabolic diseases (including diabetes); renal dysfunction; hemoglobinopathies; immune deficiency diseases (including HIV infection) or on-going immunosuppressive therapy.
* Currently pregnant; nursing mothers; or planning a pregnancy within one month of vaccination.
* Allergy to latex, egg, or egg protein, or the antibiotics neomycin or polymyxin.
* A prior serious reaction to a vaccine, or have had Guillain-Barre syndrome.
* Received an influenza vaccine in the past.
* Received any other vaccine within one month prior to enrolment
* Are participating in another research study involving any study medication

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300
Dates: Start 2006-03; Study Completion 2007-01

PRIMARY OUTCOMES:
The percentage enhancement of the immune response to Fluvax vaccine by PCC® compared to placebo as measured by hemagglutination inhibition (HAI) titre in the serum of subjects 4 weeks after vaccination

SECONDARY OUTCOMES:
Increase in T cell cytokine expression; Decrease in incidence of respiratory tract illness, an improvement in general intestinal health, and a reduction in the severity of adverse side effects of the injection

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Penny, DSc, MD, FRACP, Principal Investigator — Good Health Solutions
Locations (1):
- Good Health Solutions, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Mohamadzadeh M, Olson S, Kalina WV, Ruthel G, Demmin GL, Warfield KL, Bavari S, Klaenhammer TR. Lactobacilli activate human dendritic cells that skew T cells toward T helper 1 polarization. Proc Natl Acad Sci U S A. 2005 Feb 22;102(8):2880-5. doi: 10.1073/pnas.0500098102. Epub 2005 Feb 14. PMID 15710900
- [Background] Prescott SL, Dunstan JA, Hale J, Breckler L, Lehmann H, Weston S, Richmond P. Clinical effects of probiotics are associated with increased interferon-gamma responses in very young children with atopic dermatitis. Clin Exp Allergy. 2005 Dec;35(12):1557-64. doi: 10.1111/j.1365-2222.2005.02376.x. PMID 16393321
- [Background] Weston S, Halbert A, Richmond P, Prescott SL. Effects of probiotics on atopic dermatitis: a randomised controlled trial. Arch Dis Child. 2005 Sep;90(9):892-7. doi: 10.1136/adc.2004.060673. Epub 2005 Apr 29. PMID 15863468
- [Background] Qi H, Denning TL, Soong L. Differential induction of interleukin-10 and interleukin-12 in dendritic cells by microbial toll-like receptor activators and skewing of T-cell cytokine profiles. Infect Immun. 2003 Jun;71(6):3337-42. doi: 10.1128/IAI.71.6.3337-3342.2003. PMID 12761116